CLINICAL TRIAL: NCT03308630
Title: Immediate Effect of Energy Alignment and Mantra on Stress Related Pain in Adolescents: Stomach Aches, Musculoskeletal Pains, and Headaches
Brief Title: Immediate Effect of Energy Alignment and Mantra on Stress Related Pain in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Hong Kong Academy of Yoga Therapy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NMP/10092
Record Dates: First submitted 2017-10-08; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Stress Related Disorder; Musculoskeletal Pain; Headache
MeSH Terms: conditions — Musculoskeletal Pain; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Energy Alignment and Mantra (Experimental)
  Interventions: Behavioral: Yoga based Energy Alignment and Mantra

INTERVENTIONS:
Behavioral: Yoga based Energy Alignment and Mantra — Yoga intervention was based on the concept that there is not just a physical body, but a "subtle energy" body can be bound with residue of stress, unprocessed emotions, and excess mental energy. Using Yoga based practices combined with Mantra chants, Music and energy alignments poses, stress induced pain can be alleviated.

SUMMARY:
Psychiatrists have expressed concern at the emergence of education as a serious source of stress for school-going children - causing high incidence of deaths by suicide. Many adolescents in India are referred to hospital psychiatric units for school-related distress - exhibiting symptoms of depression, high anxiety, frequent school refusal, phobia, physical complaints, irritability, weeping spells, and decreased interest in school work. Previous studies have found significant anxiety, distress, depression, worn outs and severe impact of psychological factors on the performances of dental, engineering and medical student. But students preparing for competitive exams have not been studied yet.

Current study reports the scientific evidence of immediate effect of yoga based techniques combined with music and Vedic chants on adolescents preparing for competitive exams.

ELIGIBILITY:
Inclusion Criteria:

* All adolescents enrolled at the participating centers and that agree to sign informed consent.

Exclusion Criteria:

* not agreement to sign the informed consent

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 218 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Self reported Stress | 2 Weeks
  Stress level on the scale of 1-10 was reported before the intervention and after 2 week of practice

SECONDARY OUTCOMES:
Change in Musculo-skeleton Pain measured on VAS | 2 weeks
  VAS at the beginning and end of the 2 week of intervention
Change in Headache severity on VAS | 2 weeks
  VAS at the beginning and end of the 2 week of study intervention
Change in Stomach pain on VAS | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Meghwal, Principal Investigator — Hong Kong Academy of yoga therapy, Hong Kong; Neha Sharma, PhD, Study Director — Warwick Research Services; Puneet Sharma, Study Chair — NMP Medical Research Institute, India
Locations (1):
- NMP Medical Research Institute, Bikaner, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided